CLINICAL TRIAL: NCT04435444
Title: Pilot of a Meaning-Centered Intervention for Muslims Undergoing Treatment for Stage III or IV Cancer
Brief Title: Meaning-Centered Intervention for Muslim Patients Who Are Being Treated for Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-018
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancer
Keywords: Meaning-Centered Intervention; Masterful intervention; 20-018

STUDY DESIGN:
Intervention Model Description: 2-group randomized controlled trial (RCT). Using a consecutive patient sampling scheme, we will randomize Muslim patients with stage III or IV cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masterful supportive care (Experimental): This intervention uses teachings, discussions, and exercises about personal experiences that focus on specific topics related to meaning and cancer. For example, we may discuss what is meaningful in your life, how you identify yourself before and after cancer, and your hopes for the future. The Masterful intervention is available in both English and Arabic, and it will be delivered by a trained bilingual member of the study team. It includes 3 weekly (or at participant's preference) 1-hour sessions with a member of the study team. The sessions for either the treatment or the control arm will take place in-person in a private room at MSKCC or via teleconference, depending on the patients preference. Meeting one-on-one with an interventionist was feasible in our pilot study and will enhance relationship-building between interventionist and patient. Participants will have the option to meet with the interventionist via teleconference in order to reduce in-person contact burden.
  Interventions: Other: Masterful supportive care
- Attention control supportive care (Active Comparator): This intervention uses the American Cancer Society's patient education materials. These sessions will include discussions about managing a self-identified current problem in your life. The attention control supportive care intervention is available in both English and Arabic, and it will be delivered by a trained bilingual member of the study team. It includes 3 weekly (or at participant's preference) 1-hour sessions with a member of the study team. The sessions for either the treatment or the control arm will take place in-person in a private room at MSKCC or via teleconference, depending on the patients preference. Meeting one-on-one with an interventionist was feasible in our pilot study and will enhance relationship-building between interventionist and patient. Participants will have the option to meet with the interventionist via teleconference in order to reduce in-person contact burden.
  Interventions: Other: Attention control supportive care

INTERVENTIONS:
Other: Masterful supportive care — Three study questionnaires:
  Functional Assessment of Cancer Therapy-General* (FACT-G), Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being* (FACIT-Sp) Memorial Symptom Assessment Scale Short Form* (MSAS-SF)
  Arms: Masterful supportive care
Other: Attention control supportive care — Three study questionnaires:
  Functional Assessment of Cancer Therapy-General* (FACT-G), Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being* (FACIT-Sp) Memorial Symptom Assessment Scale Short Form* (MSAS-SF)
  Arms: Attention control supportive care

SUMMARY:
This study will compare the effectiveness of the Masterful supportive care intervention with that of the non-faith-based active control supportive care intervention, which uses the American Cancer Society's patient education materials, for Muslim patients who have advanced cancers.

All 3 sessions may occur within one week or over multiple weeks (nonconsecutively), depending on the participants preference. The participant will have up to 12 weeks from recruitment to complete all sessions and follow up surveys.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* identify, either as self-report or on the MSKCC EMR, as Muslim
* are in treatment including surveillance, for a confirmed diagnosis of stage III or IV cancer (solid or liquid) as per clinician or pathology report
* have an estimated life expectancy of at least 6 months, as determined by their primary oncologist
* are cognitively intact (oncologist's clinical impression or judgement of study staff)
* able to speak and read English or Arabic (self-reported preference or on the MSKCC EMR system).
* To assess English proficiency, participants will be asked two questions: (1) the Census limited English proficient item "How well do you speak English?" with response options "Not at all, Not well, Well, or Very well" and (2) "What is your preferred language for healthcare?"
* Participants who are eligible for the study and are fluent in English will be identified by the response "Very well" to the 1st question and a response indicating English as the preferred language for healthcare.

Exclusion Criteria:

* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation
* patients diagnosed with primary brain tumors as per clinician report, as they may have difficulty completing the intervention and answering the questionnaires
* undergoing hematopoietic stem cell transplantation (HSCT) as per clinican report or the EMR
* currently in psychotherapeutic treatment. Symptoms of anxiety and depression are common among patients with stage III or IV cancer. Antidepressants, anxiolytics, and other psychotropic medications do not diminish the effects of psychotherapy; thus we will not exclude patients who are being treated with these medications, as long as they are not in psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
number of enrolled participants completing at least one psychotherapy session out of the planned three. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm